CLINICAL TRIAL: NCT01483573
Title: Effect of Hamstring Stretching and Neural Mobilization on Range of Motion and Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment over time
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0120100079
Record Dates: First submitted 2010-10-07; First posted 2011-12-01 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain
Keywords: low back pain; straight leg raise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- straight leg raise (Experimental): stretch the muscle
  Interventions: Other: straight leg raise
- neural mobilization (Experimental): stretch the nerve
  Interventions: Other: neural mobilization

INTERVENTIONS:
Other: neural mobilization — stretch the nerve
  Arms: neural mobilization
Other: straight leg raise — stretch the hamstring
  Other Names: hamstring stretching
  Arms: straight leg raise

SUMMARY:
This study was designed to answer 3 primary research questions:

1. In adults with low back pain, reduced SLR ROM (Range of Motion) and a positive sensitized SLR (Straight leg raise) test, does neurodynamic mobilization result in greater SLR ROM, pain reduction and perceived improvement than muscle stretching?
2. In adults with low back pain, reduced SLR ROM and a negative sensitized SLR test, does muscle stretching result in greater SLR ROM, pain reduction and perceived improvement than neurodynamic mobilization?
3. In adults with low back and reduced SLR, does neurodynamic mobilization or muscle stretching result in greater SLR ROM, pain reduction and perceived improvement irrespective of the outcome of SLR sensitization?

The research hypotheses are threefold:

1. Subjects determined to have nerve-related pain and ROM restrictions by a positive sensitized SLR test would benefit more from neurodynamic mobilization than muscle stretching.
2. Subjects determined to have muscle-related pain and ROM restrictions by a negative sensitized SLR test would benefit more from muscle stretching than neurodynamic mobilization.
3. Subjects would benefit the same from muscle stretching and neurodynamic mobilization when not matched on the outcome of the SLR sensitization.

DETAILED DESCRIPTION:
Potential subjects will sign an informed consent and be evaluated for inclusion in the study. Subjects meeting the inclusion criteria will be asked to complete a form asking questions regarding their demographics, pain history and symptomatology. The form will also include a numeric pain rating scale to determine pain severity, and a standardized questionnaire commonly used in back pain research (i.e., the Modified Oswestry Disability Index). Subjects will then be evaluated for SLR range of motion on the side with the least amount of SLR range of motion using a bubble inclinometer.

Subjects will then be randomly assigned to receive a treatment to address hamstring length or a treatment to address sciatic nerve restrictions. A second researcher who is blinded to the results of the data obtained pre-treatment will administer the treatment. Hamstring stretching will consist of positioning the subject's hip in flexion and knee in extension, and holding this position for 30 seconds. This treatment will be repeated 5 times. Nerve mobilization will consist of either momentarily positioning the hip in flexion, the knee in extension and the ankle in dorsiflexion, and then moving the ankle in and out of dorsiflexion at a rate of about 1 - 2 movements per second (theoretically, this should stretch the nerve), or moving the lower leg such that it is first positioned into hip extension and ankle dorsiflexion, and then into hip flexion and ankle plantarflexion (theoretically, this should glide the nerve in its sheath). The choice of technique will be made by the treating therapist. Both treatments should take approximately 4 minutes to complete.

Following this intervention, subjects will be re-evaluated for SLR range of motion using a bubble inclinometer by the same researcher who collected the pre-treatment data. During the next visit to physical therapy, this researcher will re-evaluate subjects SLR range of motion, as previously described; and pain, by the numeric pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to physical therapy for low back pain with limitations in hamstring range of motion on the painful side

Exclusion Criteria:

* Red flags

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
range of motion | within 72 hours
  Measured with a bubble inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Edmond, PT, DSc, OCS, Study Director — University of Medicine and Dentistry
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Decoster LC, Cleland J, Altieri C, Russell P. The effects of hamstring stretching on range of motion: a systematic literature review. J Orthop Sports Phys Ther. 2005 Jun;35(6):377-87. doi: 10.2519/jospt.2005.35.6.377. PMID 16001909
- [Background] Coppieters MW, Butler DS. Do 'sliders' slide and 'tensioners' tension? An analysis of neurodynamic techniques and considerations regarding their application. Man Ther. 2008 Jun;13(3):213-21. doi: 10.1016/j.math.2006.12.008. Epub 2007 Mar 30. PMID 17398140
- [Background] Schafer A, Hall T, Briffa K. Classification of low back-related leg pain--a proposed patho-mechanism-based approach. Man Ther. 2009 Apr;14(2):222-30. doi: 10.1016/j.math.2007.10.003. Epub 2007 Dec 31. PMID 18165145
- [Background] Schafer A, Hall T, Muller G, Briffa K. Outcomes differ between subgroups of patients with low back and leg pain following neural manual therapy: a prospective cohort study. Eur Spine J. 2011 Mar;20(3):482-90. doi: 10.1007/s00586-010-1632-2. Epub 2010 Dec 1. PMID 21116662
- [Background] Boyd BS, Wanek L, Gray AT, Topp KS. Mechanosensitivity of the lower extremity nervous system during straight-leg raise neurodynamic testing in healthy individuals. J Orthop Sports Phys Ther. 2009 Nov;39(11):780-90. doi: 10.2519/jospt.2009.3002. PMID 19881004